CLINICAL TRIAL: NCT06322680
Title: The Impact of External Drainage of the Main Pancreatic Duct and Common Bile Duct on Pancreatic Fistula Following Pancreaticoduodenectomy: A Multi-center Prospective Randomized Controlled Phase Clinical Trial
Brief Title: Impact of External Drainage of the Main Pancreatic Duct and Common Bile Duct on Pancreatic Fistula Following Pancreaticoduodenectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Huadong Hospital (Other); RenJi Hospital (Other); The First People's Hospital of Yunnan (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-03
Record Dates: First submitted 2024-03-08; First posted 2024-03-21 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-05

CONDITIONS: Pancreaticoduodenectomy
Keywords: Pancreaticoduodenectomy; postoperative pancreatic fistula; delayed gastric emptying; post-pancreatectomy hemorrhage; biliary leakage
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: Prospective, Multicenter, Controlled, Superiority Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main pancreatic duct and biliary duct external drainage (Experimental): Pancreaticojejunostomy:
  Assess pancreatic texture and duct diameter, preparing a 2 cm pancreatic remnant, and securing it to the jejunum's muscular layer using 3-0 prolene for U-shaped anastomosis. A patented drainage tube is inserted into the jejunum for effective drainage. Anastomoses are performed with 4-0 prolene between the pancreatic duct and jejunal mucosa, both posteriorly and anteriorly, with additional reinforcement at the pancreas and jejunum's anterior walls. A Fr6 silicone tube is placed in the distal jejunal remnant and secured.
  The drainage system, featuring a one-way valve, connects the internal and external silicone tubes to a drainage bag.
  Choledochojejunostomy:
  The common bile duct's diameter is noted, and an opening in the jejunum is made for hepatobiliary tract formation with 4-0 absorbable sutures. A Fr10 silicone tube is inserted into the afferent limb and secured. This tube, too, connects to the external drainage system with a one-way valve.
  Interventions: Procedure: Main pancreatic duct and biliary duct external drainage
- Main pancreatic duct and biliary duct internal drainage (Experimental): Pancreaticojejunostomy:
  Assess the pancreatic texture and pancreatic duct diameter, and reserve the length of the pancreatic remnant to about 1.5 cm. Open the transverse mesocolon and bring the distal small intestinal remnant to the side of the pancreatic remnant. Perform a 2 cm side-to-side pancreaticojejunostomy with an invagination technique. Use a simple full-layer suturing method, 4-0 PDS plus continuous suturing, insert a plastic strip into the pancreatic duct, and fix the pancreatic duct stent with 3/0 Vicryl.
  Choledochojejunostomy:
  Record the diameter of the common bile duct, about 10 cm away from the pancreaticojejunostomy, and open the jejunum. Form the hepatobiliary tract and perform interrupted anastomosis with 4-0 absorbable sutures.
  Interventions: Procedure: Main pancreatic duct and biliary duct internal drainage

INTERVENTIONS:
Procedure: Main pancreatic duct and biliary duct external drainage — Pancreaticojejunostomy:
  Assess pancreatic texture and duct diameter, preparing a 2 cm pancreatic remnant, and securing it to the jejunum's muscular layer using 3-0 prolene for U-shaped anastomosis. A patented drainage tube is inserted into the jejunum for effective drainage. Anastomoses are performed with 4-0 prolene between the pancreatic duct and jejunal mucosa, both posteriorly and anteriorly, with additional reinforcement at the pancreas and jejunum's anterior walls. A Fr6 silicone tube is placed in the distal jejunal remnant and secured.
  The drainage system, featuring a one-way valve, connects the internal and external silicone tubes to a drainage bag.
  Choledochojejunostomy:
  The common bile duct's diameter is noted, and an opening in the jejunum is made for hepatobiliary tract formation with 4-0 absorbable sutures. A Fr10 silicone tube is inserted into the afferent limb and secured. This tube, too, connects to the external drainage system with a one-way valve.
  Arms: Main pancreatic duct and biliary duct external drainage
Procedure: Main pancreatic duct and biliary duct internal drainage — Pancreaticojejunostomy:
  Assess the pancreatic texture and pancreatic duct diameter, and reserve the length of the pancreatic remnant to about 1.5 cm. Open the transverse mesocolon and bring the distal small intestinal remnant to the side of the pancreatic remnant. Perform a 2 cm side-to-side pancreaticojejunostomy with an invagination technique. Use a simple full-layer suturing method, 4-0 PDS plus continuous suturing, insert a plastic strip into the pancreatic duct, and fix the pancreatic duct stent with 3/0 Vicryl.
  Choledochojejunostomy:
  Record the diameter of the common bile duct, about 10 cm away from the pancreaticojejunostomy, and open the jejunum. Form the hepatobiliary tract and perform interrupted anastomosis with 4-0 absorbable sutures.
  Arms: Main pancreatic duct and biliary duct internal drainage

SUMMARY:
Pancreaticoduodenectomy (PD) is the standard treatment for tumors of the pancreatic head, distal bile duct, duodenum, and ampulla of Vater. With advances in surgical experience and instrumentation, the mortality rate of PD has decreased to below 5% in high-volume pancreatic centers. However, the postoperative complication rate remains high at 25%-50%, limiting the development and application of PD.

The main postoperative complications of PD are postoperative pancreatic fistula (POPF), delayed gastric emptying (DGE), post-pancreatectomy hemorrhage (PPH), and biliary leakage (BL). POPF, BL, and the subsequent abdominal infection, PPH, etc. are the main causes of death during hospitalization. Even in large, relatively mature pancreatic centers, the incidence of POPF remains as high as 10%-40%. In recent years, various methods have been used to prevent and treat POPF and BL after PD, such as pancreatic duct stent external drainage and external biliary drainage.

To date, there have been many studies by domestic and foreign scholars on the advantages and disadvantages of biliary and pancreatic duct external drainage versus internal drainage in PD in terms of perioperative POPF incidence, mortality rate, etc., but the research results are not consistent. Overall, pancreatic duct stent external drainage is only recommended for patients with a high risk of pancreatic fistula during PD. Currently, there have been a few relevant studies exploring and verifying the preventive effect of pancreatic duct stent external drainage on pancreatic fistula in patients with high risk of pancreatic fistula. For example, a retrospective study of 98 patients with soft pancreatic parenchyma by Teruyuki Usub et al. found that there was no significant difference between groups with and without pancreatic duct stent in preventing pancreatic fistula. However, due to the low level of evidence, only a few risk factors such as pancreatic texture and pancreatic duct diameter were included, and the risk of POPF was not systematically evaluated. Further clinical exploration and verification are needed. In 2013, Mark P Callery et al. proposed a pancreatic fistula risk score (The fistula risk score, FRS) based on the pancreatic fistula standard defined by the International Pancreatic Fistula Study Group, which included pancreatic texture, pathological type, pancreatic duct diameter, and intraoperative blood loss. This model can be used to systematically and quantitatively evaluate the risk of POPF. Previous studies did not have a clear stratification for patients undergoing pancreatic duct stent external drainage, which may have included too many patients with a low risk of pancreatic fistula, resulting in inaccurate results. Therefore, it is necessary to re-evaluate the effectiveness of pancreatic duct stent external drainage in preventing clinically relevant pancreatic fistula based on stratification of pancreatic fistula risk and disease type. At the same time, pancreatic juice contains a variety of digestive enzymes, of which pancreatic lipase, trypsin, and chymotrypsin all need to be activated by bile to play a role in digesting and decomposing fat and protein. Theoretically, biliary and pancreatic juice diversion may be able to reduce the incidence of pancreatic fistula and its related complications in PD patients.

Thus, the investigators design the present study to evaluate the impact of main pancreatic duct and biliary duct external drainage on postoperative complication, especially POPF.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is the standard treatment for tumors of the pancreatic head, distal bile duct, duodenum, and ampulla of Vater. With advances in surgical experience and instrumentation, the mortality rate of PD has decreased to below 5% in high-volume pancreatic centers. However, the postoperative complication rate remains high at 25%-50%, limiting the development and application of PD.

The main postoperative complications of PD are postoperative pancreatic fistula (POPF), delayed gastric emptying (DGE), post-pancreatectomy hemorrhage (PPH), and biliary leakage (BL). POPF, BL, and the subsequent abdominal infection, PPH, etc. are the main causes of death during hospitalization. Even in large, relatively mature pancreatic centers, the incidence of POPF remains as high as 10%-40%. In recent years, various methods have been used to prevent and treat POPF and BL after PD, such as pancreatic duct stent external drainage and external biliary drainage.

To date, there have been many studies by domestic and foreign scholars on the advantages and disadvantages of biliary and pancreatic duct external drainage versus internal drainage in PD in terms of perioperative POPF incidence, mortality rate, etc., but the research results are not consistent. Overall, pancreatic duct stent external drainage is only recommended for patients with a high risk of pancreatic fistula during PD. Currently, there have been a few relevant studies exploring and verifying the preventive effect of pancreatic duct stent external drainage on pancreatic fistula in patients with high risk of pancreatic fistula. For example, a retrospective study of 98 patients with soft pancreatic parenchyma by Teruyuki Usub et al. found that there was no significant difference between groups with and without pancreatic duct stent in preventing pancreatic fistula. However, due to the low level of evidence, only a few risk factors such as pancreatic texture and pancreatic duct diameter were included, and the risk of POPF was not systematically evaluated. Further clinical exploration and verification are needed. In 2013, Mark P Callery et al. proposed a pancreatic fistula risk score (The fistula risk score, FRS) based on the pancreatic fistula standard defined by the International Pancreatic Fistula Study Group, which included pancreatic texture, pathological type, pancreatic duct diameter, and intraoperative blood loss. This model can be used to systematically and quantitatively evaluate the risk of POPF. Previous studies did not have a clear stratification for patients undergoing pancreatic duct stent external drainage, which may have included too many patients with a low risk of pancreatic fistula, resulting in inaccurate results. Therefore, it is necessary to re-evaluate the effectiveness of pancreatic duct stent external drainage in preventing clinically relevant pancreatic fistula based on stratification of pancreatic fistula risk and disease type. At the same time, pancreatic juice contains a variety of digestive enzymes, of which pancreatic lipase, trypsin, and chymotrypsin all need to be activated by bile to play a role in digesting and decomposing fat and protein. Theoretically, biliary and pancreatic juice diversion may be able to reduce the incidence of pancreatic fistula and its related complications in PD patients.

Thus, the investigators design the present study to evaluate the impact of main pancreatic duct and biliary duct external drainage on postoperative complication, especially POPF.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 80 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Life expectancy ≥12 weeks and ASA score ≤2.
* Based on clinical symptoms, imaging examinations, tumor markers, and other auxiliary examinations, the clinical diagnosis includes but is not limited to tumors of the pancreatic head, ampulla of Vater, duodenum, and distal common bile duct, requiring pancreaticoduodenectomy.
* No serious dysfunction in blood system, heart, lung function, or autoimmune system (refer to the respective diagnostic criteria)
* White blood cell (WBC) ≥ 3 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets (PLT) ≥ 100 × 109/L; Hemoglobin (Hgb) ≥ 90 g/L
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal (ULN); Total bilirubin (TBIL) ≤ ULN; Creatinine (CRE) ≤ 1.5 × ULN
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 × ULN
* Able to comply with research visit plans and other protocol requirements.
* With intermediate or high risk of postoperative pancreatic fistula (POPF) according to alternative fistula risk scoring system (A-FRS)

Exclusion Criteria:

* Cancer in late stage including distant organ metastasis (liver, lung, peritoneum), metastasis to the hilar bile duct and hepatic duct, extensive metastasis to the hepatic portal lymph nodes, tumor invasion of the superior mesenteric artery, celiac trunk, inferior vena cava, or abdominal aorta.
* Heart Failure: Congestive heart failure with New York Heart Association (NYHA) heart function classification of 3 or 4.
* Uncontrolled Hypertension:
* Renal Failure: Renal failure or insufficiency requiring hemodialysis or peritoneal dialysis.
* Active Infection: Serious active clinical infection (> Grade 2, NCI-CTCAE version 4.0).
* Pregnancy or Lactation: Pregnant or lactating women.
* Major Surgery: Patients who have undergone major surgery within 4 weeks of starting the trial or have not recovered from the side effects of such surgery.
* Other Malignancies: Combined with other malignant tumors (patients who have been cured 3 years ago can be included).
* Upper Gastrointestinal Bleeding: Excluding patients with upper gastrointestinal bleeding within 4 weeks before surgery or with a clear tendency of gastrointestinal bleeding that cannot be corrected by active medical treatment.
* Poor Compliance: Poor compliance, unable or unwilling to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of clinically relevant postoperative pancreatic fistula (B/C grade fistula) within 90 days after surgery | From date of surgery to postoperative day 90.
  To evaluate the incidence of clinically relevant postoperative pancreatic fistula (B/C grade fistula) within 90 days after surgery. Medical record, outpatient visit, phone interview.

SECONDARY OUTCOMES:
Surgical Complications: Incidence and grading of complications within 90 days after surgery | From date of surgery to postoperative day 90.
  To evaluate the incidence of surgical complications mentioned above within 90 days after surgery. Medical record, outpatient visit, phone interview.
  Incidence and grading of complications within 90 days after surgery:
  Pancreatic fistula (A/B/C grade) Biliary fistula Chylothorax Gastrointestinal/intestinal anastomotic fistula Postoperative pancreatic hemorrhage Gastric emptying disorders Intra-abdominal infection Lower extremity deep vein thrombosis Pulmonary embolism Myocardial infarction Cerebral infarction Incisional complications
Surgical Complications: Clavien-Dindo classification | From date of surgery to postoperative day 90.
  To evaluate the Clavien-Dindo classification within 90 days after surgery. Medical record, outpatient visit, phone interview.
Surgical Complications: Mortality rate | From date of surgery to postoperative day 90.
  To evaluate the rate mentioned above within 90 days after surgery. Medical record, outpatient visit, phone interview
Surgical Complications: reoperation rate | From date of surgery to postoperative day 90.
  To evaluate the rate mentioned above within 90 days after surgery. Medical record, outpatient visit, phone interview
Surgical Complications: readmission rate | From date of surgery to postoperative day 90.
  To evaluate the rate mentioned above within 90 days after surgery. Medical record, outpatient visit, phone interview
Surgical Complications: rate of digital subtraction angiography for postoperative pancreatic hemorrhage | From date of surgery to postoperative day 90.
  To evaluate the rate mentioned above within 90 days after surgery. Medical record, outpatient visit, phone interview
Surgical Complications: Total cost of perioperative treatment | From date of surgery to the date of discharge, an average of 2 weeks.
  To evaluate the total cost of perioperative treatment. Medical record.
Surgical Complications: Length of hospital stay | From date of surgery to the date of discharge, an average of 2 weeks.
  To evaluate the length of hospital stay. Medical record.
Adjuvant treatment: Proportion of patients with delayed adjuvant treatment (≥12 weeks) due to complications such as pancreatic fistula after surgery | From date of surgery to the date of starting adjuvant treatment, an average of 1 month.
  To evaluate proportion of patients with delayed adjuvant treatment (≥12 weeks) due to complications such as pancreatic fistula after surgery. Medical record, outpatient visit, phone interview.
Adjuvant treatment: Interval between the start of adjuvant treatment and surgery | From date of surgery to the date of starting adjuvant treatment, an average of 1 month.
  To evaluate the interval between the start of adjuvant treatment and surgery. Medical record, outpatient visit, phone interview.
Long-term survival related to malignant tumors: Overall survival (OS) | From date of surgery until the date of death from any cause, assessed 3 months thereafter up to 60 months
  Overall survival after surgery. To evaluate the overall survival of patients after surgery. Outpatient visit, phone interview.
Long-term survival related to malignant tumors: Disease-free survival (DFS) | From date of surgery until the date of death from any cause, assessed 3 months thereafter up to 60 months
  Disease-free survival after surgery. To evaluate the disease-free survival of patients after surgery. Outpatient visit, phone interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang WQ, Xu YL, Tang LH, He JY, Li Y, Liang F, Zhang YM, Gan W, Xu HX, Zhang L, Wu WC, Shi CY, Jin Y, Jiang CY, Wang Z, He M, Wang XA, Qiu YD, Liu L. Impact of external drainage of the main pancreatic duct and common bile duct on postoperative pancreatic fistula following pancreatoduodenectomy: protocol for a multicentre randomized clinical trial. BJS Open. 2025 Oct 30;9(6):zraf130. doi: 10.1093/bjsopen/zraf130. PMID 41189489